CLINICAL TRIAL: NCT07054970
Title: A Phase 1, Randomized, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety and Immunogenicity of CT-P55, EU-approved Cosentyx and US-licensed Cosentyx in Healthy Male Subjects
Brief Title: To Compare the Pharmacokinetics, Safety and Immunogenicity of CT-P55 and Cosentyx in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CT-P55 1.1
Record Dates: First submitted 2025-06-22; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CT-P55 (Experimental): a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: CT-P55
- US-licensed Cosentyx (Active Comparator): a single SC injection via PFS
  Interventions: Biological: US-licensed Cosentyx
- EU-approved Cosentyx (Active Comparator): a single SC injection via PFS
  Interventions: Biological: EU-approved Cosentyx

INTERVENTIONS:
Biological: CT-P55 — 150 mg in 1.0 mL, administered as a single SC injection via PFS
  Arms: CT-P55
Biological: US-licensed Cosentyx — 150 mg in 1.0 mL, administered as a single SC injection via PFS
  Arms: US-licensed Cosentyx
Biological: EU-approved Cosentyx — 150 mg in 1.0 mL, administered as a single SC injection via PFS
  Arms: EU-approved Cosentyx

SUMMARY:
This is a Phase 1, Randomized, Double-blind, three-arm, Parallel group, Single-dose Study to Compare the Pharmacokinetics, Safety and immunogenicity of CT-P55, EU-approved Cosentyx and US-licensed Cosentyx in Healthy male Subjects

DETAILED DESCRIPTION:
CT-P55, containing the active ingredient secukinumab, is being developed by CELLTRION, Inc. as a proposed biosimilar to the reference product, Cosentyx. In this study, Pharmacokinetics, Safety and Immunogenicity of CT-P55, EU-approved Cosentyx and US-licensed Cosentyx were evaluated in Healthy Male Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, both inclusive.
* Body weight between 50.0 kg and 90.0 kg (both inclusive), and Body Mass Index (BMI) between 18.5 and 29.9 kg/m2 (both inclusive), when rounded to the nearest tenth.

Exclusion Criteria:

* A medical history and/or condition that is considered significant
* Clinically significant allergic reactions, hypersensitivity
* History or current infection of human immunodeficiency virus, hepatitis B virus, hepatitis C virus or syphilis
* Active or latent Tuberculosis
* History of malignancy
* Previous monoclonal antibody or fusion protein treatment, or current use of any biologics
* Planning to be father a child or donate sperm within 22 weeks period following study drug administration.
* Undergone treatment with an investigational drug or participated in another clinical trial within 12weeks or 5 half-lives (whichever is longer)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) similarity demonstration in terms of area under the concentration-time curve (AUC) from time zero to infinity (AUC0-inf) | Day 155
  Demonstrate PK similarity in terms of area under the concentration-time curve (AUC) from time zero to infinity (AUC0-inf) of CT-P55, European Union (EU)-approved Cosentyx and United States (US)-licensed Cosentyx in healthy male subjects. The similarity of PK will be concluded if the 90% Cls for the ratios of geometric means of the comparison are entirely contained within the equivalence margin of 80% to 125% for AUC0-inf.
PK similarity demonstration in terms of maximum serum concentration (Cmax) | Day 155
  Demonstrate PK similarity in terms of Cmax of CT-P55, EU-approved Cosentyx and US-licensed Cosentyx in healthy male subjects up to Day 155. The similarity of PK will be concluded if the 90% Cls for the ratios of geometric means of the comparison are entirely contained within the equivalence margin of 80% to 125% for Cmax.

SECONDARY OUTCOMES:
Evaluate additional PK in terms of AUC from time zero to the last quantifiable concentration (AUC0-last) | Day 155
Evaluate additional PK in terms of Time to Cmax (Tmax) | Day155
Evaluate additional PK in terms of Apparent volume of distribution during the terminal phase after non-intravenous administration (Vz/F) | Day 155
Evaluate additional PK in terms of Terminal elimination rate constant (λz) | Day155
Evaluate additional PK in terms of Terminal elimination half-life (t1/2) | Day 155
Evaluate additional PK in terms of Apparent total body clearance (CL/F) | Day155
Evaluate additional PK in terms of Percentage of the area extrapolated for calculation of AUC0-inf (%AUCextrap) | Day 155
Evaluate safety in terms of treatment-emergent adverse events (TEAEs) of CT-P55 as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. | Day 155

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Hasunuma, Principal Investigator — Kitasato University Kitasato Institute Hospital
Locations (4):
- Japan (4):
  - Yokohama Minoru Clinic, Yokohama, Kanagawa
  - SOUSEIKAI Nishikumamoto Hospital, Kumamoto, Kumamoto
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasunuma T, Yagi M, Nakamichi N, Blauvelt A, Thaci D, Suh J, Cha J, Noh I, Lee E, Papp KA. Pharmacokinetics and safety of candidate biosimilar CTP55 versus reference secukinumab: a three-arm, randomized, double-blinded, single-dose, multicenter, phase I study. Expert Opin Investig Drugs. 2026 Feb 10. doi: 10.1080/13543784.2026.2628208. Online ahead of print. PMID 41665131